CLINICAL TRIAL: NCT04169880
Title: Effects of High Intensity Laser Therapy (HILT) in Patients With Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Collaborators: Scientific Research Projects (Unknown)
Responsible Party: Principal Investigator, Seda Paskal, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1495-GOA 2015/23-30
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Subacromial impingement syndrome; High Intensity Laser Therapy; Laser Therapy; Shoulder Pain
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Our study is a parallel group randomised comparison trial comparing two interventions with a 1:1 ratio.
Who Masked: Participant
Masking Description: The author who did not perform evaluation or treatment of the patients assessed participants for eligibility and assigned them to one of the two groups; HILT (n=15) and HILT&Exercise (n=15) (Figure 1) by a computerized random number generator (Random.org; Randomness and Integrity Services Ltd, Dublin, Ireland; httpp://www.random.org). Participants did not know there were two groups and which group they were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HILT Group (Experimental): HILT Group (n=15)
  Interventions: Device: HILT
- HILT & EXERCISE Group (Experimental): HILT&Exercise Group (n=15)
  Interventions: Combination Product: HILT & EXERCISE

INTERVENTIONS:
Device: HILT — HILT will be performed with BTL 6000 High Intensity Laser (London, UK) which is a therapeutic non-invasive neodymium: yttrium aluminum garnet laser that has a pulsating waveform and 1064 nm wavelength, 12 Watt maximum power and has the ability to penetrate 12 cm.
  Other Names: BTL 6000 High Intensity Laser (London, UK)
  Arms: HILT Group
Combination Product: HILT & EXERCISE — HILT&Exercise group will receive exercise therapy right after they receive HILT. Both groups will receive treatment for 3 days a week, on alternate days and totally 10 sessions. Patients will be asked not to use analgesic medication throughout the treatment period.
  Arms: HILT & EXERCISE Group

SUMMARY:
The aim of this study is to determine the effects of high intensity laser therapy (HILT) in patients with subacromial impingement syndrome (SIS). This study aims to compare the effects of HILT alone and HILT and therapeutic exercise combination on shoulder pain, ROM, joint position sense (JPS), muscle strength and function.The investigators hypothesized that shoulder pain, ROM, JPS, muscle strength and functionality would improve with both treatments but that HILT combined with exercise would result in better outcomes than HILT alone.

DETAILED DESCRIPTION:
30 patients with SIS will be randomized into two groups. Pain intensity will be assessed with visual analogue scale (VAS), pain-free and normal range of motion (ROM) with goniometer, joint position sense (JPS) with inclinometer, muscle strenght with hand-held dynamometer, and shoulder functionality with Constant Murley Score (CMS) and Shoulder Pain and Disability Index (SPADI) in a pretest-posttest design. HILT Group (n=15) will receive only HILT for 10 sessions, 3 days a week on alternate days. HILT& Exercise Group (n=15) will receive exercise treatment in addition to HILT for the same duration of time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as SIS (≥3 positive of 5 impingement tests: Neer's sign, Hawkins and Kennedy, Empty Can, painful arc of abduction and external rotation resistance tests)
* No history of shoulder injury and/or shoulder symptoms requiring treatment other than SIS for the last 1 year
* Shoulder pain less than 7/10 of Visual Analogue Scale
* Being able to elevate the shoulder over 140 degrees

Exclusion Criteria:

* History of upper extremity fracture, shoulder surgery
* Frozen shoulder
* Full-thickness rotator cuff (RC) tear
* Shoulder instability, systemic musculoskeletal disease
* Shoulder pain with cervical spine motion,
* Having any of the contraindications of HILT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05-05 (Actual); Primary Completion 2016-01-06 (Actual); Study Completion 2016-05-27 (Actual)

PRIMARY OUTCOMES:
Pain Evaluation:Visual Analogue Scale (VAS) | 4 weeks
  Rest and activity pain of the shoulder will be measured on a 10-cm VAS ranging from 0 (no pain) to 10 (worst pain imaginable). Higher scores mean worse outcome.
Shoulder Range of Motion Evaluation | 4 weeks
  Active and passive ROM will be evaluated with universal goniometer (Baseline®, Fabrication End Inc, New York, USA).
Pain-free Range of Motion Evaluation | 4 weeks
  Pain-free ROM will be assessed by measuring pain-free ROM for active shoulder elevation in scapular plane with universal goniometer. While sitting on a chair with back support, patients performed elevation with their thumbs pointing up. One degree below the angle where the patient first experienced pain was recorded.
Muscle Strength Evaluation | 4 weeks
  A hand-held dynamometer (HHD) (Power track II, J Tech, New York, USA) will be used to assess muscle strength. Before the evaluations test order will be randomized for lower trapezius (LT), middle trapezius (MT), upper trapezius (UT), serratus anterior (SA), supraspinatus (SupraSp), subscapularis (SubSc), infraspinatus&teres minor (IS&TM) muscles.
Shoulder Joint Position Sense (JPS) Evaluation | 4 weeks
  A bubble inclinometer (Baseline®, Fabrication End Inc, NewYork, USA) will be used to assess active shoulder JPS. The inclinometer will be attached to an elastic strip via a velcro-band and placed on proximal humerus for abduction and on wrist for rotations. Shoulder JPS in abduction direction will be evaluated while patient sitting on a chair without back support at the angle of 100°, 19 internal rotation (IR) and external rotation (ER); while patient lying supine, at the angles of 45° IR and 75° ER.
Shoulder Function and Disability Evaluation | 4 weeks
  The Turkish version of the Shoulder Pain and Disability Index (SPADI) will be used to evaluate shoulder disability level. Items in the index are presented on a numerical rating scale (0 indicates no pain/no difficulty, 10 indicates worst pain/most difficulty). Higher score indicates greater disability.
  The Turkish version of the Constant-Murley Shoulder Score (CMS) will be used to evaluate shoulder function. It is a 100-points-scale composed of pain (15 points), activities of daily living (ADL) (20 points), active ROM (40 points) and strenght (25 points) subgroups. The total score is classified as excellent (90-100), good (80-89), moderate (70-79) and weak (<70).

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Sevi Yeşilyaprak, Assoc. Prof. PT., Principal Investigator — Dokuz Eylul University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pekyavas NO, Baltaci G. Short-term effects of high-intensity laser therapy, manual therapy, and Kinesio taping in patients with subacromial impingement syndrome. Lasers Med Sci. 2016 Aug;31(6):1133-41. doi: 10.1007/s10103-016-1963-2. Epub 2016 May 25. PMID 27220527
- [Background] Clark P, Lavielle P, Martinez H. Learning from pain scales: patient perspective. J Rheumatol. 2003 Jul;30(7):1584-8. PMID 12858463
- [Background] Riddle DL, Rothstein JM, Lamb RL. Goniometric reliability in a clinical setting. Shoulder measurements. Phys Ther. 1987 May;67(5):668-73. doi: 10.1093/ptj/67.5.668. PMID 3575423
- [Background] Michener LA, Boardman ND, Pidcoe PE, Frith AM. Scapular muscle tests in subjects with shoulder pain and functional loss: reliability and construct validity. Phys Ther. 2005 Nov;85(11):1128-38. PMID 16253043
- [Background] Turner N, Ferguson K, Mobley BW, Riemann B, Davies G. Establishing normative data on scapulothoracic musculature using handheld dynamometry. J Sport Rehabil. 2009 Nov;18(4):502-20. doi: 10.1123/jsr.18.4.502. PMID 20108852
- [Background] Anderson VB, Wee E. Impaired joint proprioception at higher shoulder elevations in chronic rotator cuff pathology. Arch Phys Med Rehabil. 2011 Jul;92(7):1146-51. doi: 10.1016/j.apmr.2011.02.004. PMID 21704796
- [Background] Haik MN, Camargo PR, Zanca GG, Alburquerque-Sendin F, Salvini TF, Mattiello-Rosa SM. Joint position sense is not altered during shoulder medial and lateral rotations in female assembly line workers with shoulder impingement syndrome. Physiother Theory Pract. 2013 Jan;29(1):41-50. doi: 10.3109/09593985.2012.676722. Epub 2012 Apr 20. PMID 22515172
- [Background] Bumin G, Tuzun EH, Tonga E. The shoulder pain and disability index (SPADI): Cross-cultural adaptation, reliability and validity of the Turkish version. J Back Musculoskelet Rehabil. 2008;21(1): 57-62. doi: 10.3233/bmr-2008-21108.
- [Background] Celik D. Turkish version of the modified Constant-Murley score and standardized test protocol: reliability and validity. Acta Orthop Traumatol Turc. 2016;50(1):69-75. doi: 10.3944/AOTT.2016.14.0354. PMID 26854052
- [Background] Steuri R, Sattelmayer M, Elsig S, Kolly C, Tal A, Taeymans J, Hilfiker R. Effectiveness of conservative interventions including exercise, manual therapy and medical management in adults with shoulder impingement: a systematic review and meta-analysis of RCTs. Br J Sports Med. 2017 Sep;51(18):1340-1347. doi: 10.1136/bjsports-2016-096515. Epub 2017 Jun 19. PMID 28630217
- [Background] Hanratty CE, McVeigh JG, Kerr DP, Basford JR, Finch MB, Pendleton A, Sim J. The effectiveness of physiotherapy exercises in subacromial impingement syndrome: a systematic review and meta-analysis. Semin Arthritis Rheum. 2012 Dec;42(3):297-316. doi: 10.1016/j.semarthrit.2012.03.015. Epub 2012 May 18. PMID 22607807